CLINICAL TRIAL: NCT04379206
Title: Social Network Approach for Increasing Testing Coverage Among Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz Ho Kwan, Postdoctoral Fellow, Chinese University of Hong Kong
Other Study IDs: MSS324R; MSS324R (Other Grant/Funding Number: AIDS Trust Fund)
Record Dates: First submitted 2020-05-02; First posted 2020-05-07 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: HIV Infections
Keywords: men who have sex with men; self-testing; social network; agent-based model; HIV; Gamification; Neumorphism
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men who have sex with men: MSM receiving a self-test kit with optional assistance
  Interventions: Diagnostic Test: HIV self-test kit; Other: Graphical User Interface

INTERVENTIONS:
Diagnostic Test: HIV self-test kit — fingerprick and oral fluid HIV self-tests with optional on-site or hotline staff assistance
Other: Graphical User Interface — Gamification or neumorphism user interface

SUMMARY:
HIV testing is essential in shortening the time to identify a new infection, the first 90 of the UNAIDS 90-90-90 targets. However, over one-third of the men who have sex with men (MSM) had never been tested for HIV; even if they did, one-fifth had their tests done more than a year ago. Assortative mixing pattern observed in the HIV-positive MSM group shaped the transmission dynamics and could be leveraged for intervention. Barriers to access HIV testing services could, on the other hand, be hurdled by self-tests. A network approach for intervention could therefore be promising in delivering effective HIV self-tests. To experiment with such an approach, a 2-phase study was conceptualised incorporating actual network-based referred HIV self-tests and an agent-based simulation evaluating its impact. Sixty-four MSM would be recruited as seeds for promoting HIV self-tests within their network and those being referred could refer their friends for the same after passing online training. To facilitate the process, an online platform would be developed offering information, collecting informed consent, requesting HIV self-test kits, returning results, performing online training, and referring peers. Participants could opt to receive self-tests by delivery or to conduct it on-site with staff assistance. A hotline with video conferencing support would be maintained to assist those who self-test at home. They could also choose between blood and oral fluid tests. Two user interfaces, namely gamification and neumorphism, would be randomly assigned. Primary outcomes to measure are number and proportion of MSM who had never or not tested within 12 months and the associating factors, and usability of the two user interfaces. Data collected in the empirical study would be used for parameterising the agent-based simulation to evaluate the impact of the approach in increasing testing coverage and shortening time to diagnosis. Its economic assessment would also be performed to cost each new infection to be identified. The approach could be feasible and effective to be adopted for future broader implementation for peer-led HIV self-test kit or HIV prevention message distribution.

ELIGIBILITY:
Inclusion Criteria:

* male
* had sex with another male in the preceding year
* able to communicate in written Chinese or English
* normally resided in Hong Kong

Exclusion Criteria:

* prisoners
* having mental illnesses that informed consent cannot be obtained

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men who have sex with men in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
effectiveness of the approach in reaching MSM who have never or not recently tested for HIV | Through study completion, at year 2
  proportion of testers who have never or not recently tested for HIV
Usability and acceptability of two user interfaces | Through study completion, at year 2
  System Usability Scores (SUS) and proportion of testers giving a score of at least 71

SECONDARY OUTCOMES:
Determinants of key actors in the social network | Through study completion, at year 2
  Network metrics predicting important actors in the referral network
Preference of two forms of HIV self-testing | Through study completion, at year 2
  Proportion of testers favouring each form of self-testing
Effect of network-based HIV self-test promotion in controlling transmission among MSM | Through study completion, at year 2
  Number of infections identified from the agent-based model
Proportion and characteristics of promoters | Through study completion, at year 2
  Promoters are testers giving an SUS score of at least 80

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley Ho Centre for Emerging Infectious Diseases, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwan TH, Lee SS. Predictors of HIV Testing and Their Influence on PrEP Acceptance in Men Who Have Sex with Men: A Cross-Sectional Study. AIDS Behav. 2018 Apr;22(4):1150-1157. doi: 10.1007/s10461-017-1978-0. PMID 29127535
- [Background] Valente TW. Network interventions. Science. 2012 Jul 6;337(6090):49-53. doi: 10.1126/science.1217330. PMID 22767921
- [Background] Kwan TH, Lee SS. Bridging Awareness and Acceptance of Pre-Exposure Prophylaxis Among Men Who Have Sex With Men and the Need for Targeting Chemsex and HIV Testing: Cross-Sectional Survey. JMIR Public Health Surveill. 2019 Jul 3;5(3):e13083. doi: 10.2196/13083. PMID 31271148
- [Background] Cao B, Saffer AJ, Yang C, Chen H, Peng K, Pan SW, Durvasula M, Liu C, Fu H, Ong JJ, Tang W, Tucker JD. MSM Behavior Disclosure Networks and HIV Testing: An Egocentric Network Analysis Among MSM in China. AIDS Behav. 2019 May;23(5):1368-1374. doi: 10.1007/s10461-019-02404-z. PMID 30680538
- [Background] Song Y, Li X, Zhang L, Fang X, Lin X, Liu Y, Stanton B. HIV-testing behavior among young migrant men who have sex with men (MSM) in Beijing, China. AIDS Care. 2011 Feb;23(2):179-86. doi: 10.1080/09540121.2010.487088. PMID 21259130
- [Background] Philbin MM, Hirsch JS, Wilson PA, Ly AT, Giang LM, Parker RG. Structural barriers to HIV prevention among men who have sex with men (MSM) in Vietnam: Diversity, stigma, and healthcare access. PLoS One. 2018 Apr 3;13(4):e0195000. doi: 10.1371/journal.pone.0195000. eCollection 2018. PMID 29614104
- [Derived] Kwan TH, Chan DPC, Wong SY, Lee SS. Implementation Cascade of a Social Network-Based HIV Self-testing Approach for Men Who Have Sex With Men: Cross-sectional Study. J Med Internet Res. 2023 Apr 26;25:e46514. doi: 10.2196/46514. PMID 37099364
- [Derived] Kwan TH, Chan DPC, Lee SS. User Experience and Usability of Neumorphism and Gamification User Interface Designs in an HIV Self-Test Referral Program for Men Who Have Sex With Men: Prospective Open-Label Parallel-Group Randomized Controlled Trial. JMIR Serious Games. 2022 Jun 22;10(2):e35869. doi: 10.2196/35869. PMID 35731564